CLINICAL TRIAL: NCT03734198
Title: A Phase II Pilot Study to Evaluate the Safety and Efficacy of the Association of Ibrutinib and Daratumumab in Relapsed/Refractory Chronic Lymphocytic Leukemia With p53 Dysfunction. IDA53 Trial. A FILO Study.
Brief Title: Evaluation of the Safety and Efficacy of the Association of Ibrutinib and Daratumumab in Relapsed/Refractory Chronic Lymphocytic Leukemia With p53 Dysfunction
Acronym: IDA53
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDA53-FILOCLL09
Record Dates: First submitted 2018-10-23; First posted 2018-11-07 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Relapsed or Refractory Chronic Lymphocytic Leukemia
Keywords: p53 dysfunction
MeSH Terms: conditions — Recurrence; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib; daratumumab

STUDY DESIGN:
Intervention Model Description: Open label multicentre phase 2 study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ibrutinib + daratumumab (Experimental): Prephase (D-27 to D0): ibrutinib 420 mg/day
  Cycle 1 (4 weeks): ibrutinib 420 mg/day from D1 to D28 + daratumumab 8 mg/kg D1 and D2, then 16 mg/kg at D8, D15, D22.
  Cycle 2 (4 weeks): ibrutinib 420 mg/day D1 to D28 + daratumumab 16 mg/kg at D1, D8, D15 and D22.
  Cycles 3 to 6 (4 weeks) : ibrutinib 420 mg/day D1 to D28 + daratumumab 16 mg/kg at D1 and D15.
  Cycles ≥ 7 (4 weeks) : ibrutinib 420 mg/day D1 to D28 + daratumumab 16 mg/kg at D1.
  Interventions: Drug: Ibrutinib; Drug: Daratumumab

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib will be given at the fixed dose of 420 mg daily for the duration of treatment.
  Other Names: Ibrutinib treatment
Drug: Daratumumab — Daratumumab will be started 28 days after beginning of ibrutinib and will be administered at the standard dose of 16 mg/kg (divided over two days for the first infusion), then 16 mg/kg for the following infusions, weekly for 2 months, then every other week for 4 months and then once a month until progression or intolerance.
  Other Names: Daratumumab perfusion

SUMMARY:
Ibrutinib, a first-in-class Bruton Tyrosine kinase (BTK) inhibitor, has become an established treatment in relapsed/refractory chronic lymphocytic leukemia (CLL). However, despite a considerable improvement of Progression Free Survival (PFS) and Overall Survival (OS) in comparison with historical controls, the prognosis of patients with 17p deletion (del17p) remains a concern, as it is clearly much less favourable than that of patient without del17p. Again, TP53 mutations correlated to poorer prognostic in Relapsed/Refractory (R/R) CLL patients treated with ibrutinib (Brown JR et al,2018). Despite these therapeutic advances, the treatment of CLL with TP53 disruption thus remains a difficult issue that warrants evaluation of alternative treatment strategies, in particular the use of ibrutinib in combination with other agents. A body of evidence suggests that targeting the extracellular molecule CD38 might be an interesting option. CD38 is a transmembrane glycoprotein with multiple receptor and enzymatic functions. The interaction of CD38 with its ligand CD31 (also known as Platelet Endothelial Cell Adhesion Molecule (PECAM-1)) not only plays a role in the binding and the migration of leucocytes through the endothelial cells wall but also triggers the activation of intracellular pathways involved in the differentiation and activation of B cells. Previous results strongly suggest that CD38 favours the expansion of CLL clones not only directly by transducing a proliferation signal but also by directing them to anatomic sites where they find favourable conditions for proliferation and survival.

Daratumumab is a first-in-class human IgG1ĸ monoclonal antibody (mAb) that binds CD38-expressing malignant cells with high affinity. Daratumumab induces tumor cell death through multiple mechanisms such as antibody-dependent cell-mediated cytotoxicity (ADCC), complement dependent cytotoxicity (CDC), antibody-dependent cellular phagocytosis (ADCP) and induction of apoptosis (de Weers et al, 2011). Recent data show that daratumumab may also display an immunomodulatory effect through depletion of a subset of immunosuppressive CD38+ Tregs (Krejcik et al, 2016). Early-stage clinical trials found daratumumab to be safe and to display encouraging clinical activity as a single agent in relapsed/refractory multiple myeloma (MM) patients (Lockhorst et al 2016, Lonial et al, 2016). Overall response rate was 31%, with rapid (median 1 month) and durable responses in this heavily pretreated MM population. Interestingly, no patient discontinued the treatment because of drug-related adverse events. These results led to approval of daratumumab in relapsed/refractory MM in December 2015. The clinical efficacy of daratumumab along with its very favourable safety profile supports its investigation in other lymphoproliferative malignancies. In particular, the expression of CD38 in poor prognosis CLL and the key role of CD38 in CLL biology provide a basis for examining the potential of daratumumab in this disease.

In preclinical studies, (Matas-Céspedes et al, 2016; Manna et al, 2017) Daratumumab efficiently kills CLL cell lines and patient-derived CLL cells by ADCC and ADCP in vitro. Daratumumab modulates CLL-T reg levels and increase cytotoxic effector T cells.

Rationale for combining ibrutinib with daratumumab:

These data suggest that combining ibrutinib with daratumumab might have a synergistic or additive effect. Both drugs inhibit B cell receptor (BCR) signalling via two different converging pathways, i.e. BTK and CD38/ZAP70/ERK (Deaglio et al, 2007). In vitro, Manna et al have shown that daratumumab is able to modulate BCR signaling.

Interestingly, the ibrutinib /daratumumab combination significantly enhanced mitochondrial-mediated apoptosis bth in CD38 high and CD38 low CLL cells (Manna et al, 2017).

Altogether, this provides a rationale for evaluating the safety and efficacy of the association of daratumumab with ibrutinib in high-risk relapsed/refractory patients for whom the standard-of-care using ibrutinib as a single agent has demonstrated limitations in terms of long-term disease control.

Primary objective of the study: to determine the efficacy of a treatment combining daratumumab and ibrutinib in a poor risk population of relapsed CLL patients with TP53 dysfunction.

Secondary objectives of the study : to determine the safety profile of daratumumab in combination with ibrutinib in CLL patients.

Inclusion period: 24 months Treatment duration (ibrutinib + daratumumab): continuous, until disease progression or unacceptable toxicity.

Follow-up period: will begin once the subject discontinues study treatment, during 2 years.

DETAILED DESCRIPTION:
This study will take place in several periods and phases of treatment:

* Observational period of selection of 28 days maximum
* Treatment period constituted:

  * a first phase of treatment with ibrutinib alone (28 days): pre-phase,
  * a formal protocol phase during which the two study drugs (ibrutinib and daratumumab) will be used together until progression of the disease or intolerance to treatment.
* 2-year follow-up period that will begin after protocol processing has been stopped.

Selection period (before starting treatment): exams performing to verify patients' eligibility.

* Collection of the medical history,
* Clinical examination with measurement of height and weight, vital signs (temperature, pulse / heart rate, blood pressure),
* Conventional blood tests to check all the functions of the body such as kidney, liver, etc
* Viral serologies (Human Immunodeficiency Virus (HIV) and hepatitis B and C) (10 ml).
* Blood Pregnancy Test for women who may have children,
* Specific blood tests to evaluate the disease and in particular to characterize the cells of LLC (mutational profile, search for chromosomal abnormalities and analysis of residual disease rate to have a reference point before the start of treatment will be made on leukemic cells),
* CT scan (thorax, abdomen and pelvis) to accurately search for and evaluate a deep tumor syndrome (lymph nodes, spleen in particular),
* Urine examination,
* Cardiological examination with an electrocardiogram (ECG)..

Treatment period: the treatment period is divided into successive cycles of 28 days.

Before starting ibrutinib and before each daratumumab cycle, a complete clinical examination and blood work will be performed.

After 12 months of treatment, an evaluation report will be made with a complete clinical examination, a complete blood test, an urinalysis if necessary, a Computed Tomography (CT) scan, a myelogram and if necessary a marrow biopsy. Regularly after this assessment (every 6 months until the end of the study), a report will be made with clinical examination, complete blood test, ECG, CT scan and if necessary, myelogram possibly associated with a marrow biopsy if justified and not previously carried out.

After the end of the protocol treatment (progression of the disease, intolerance of the protocol treatment), a last evaluation will be carried out within 30 days after the last taking of the protocol treatment. This evaluation includes a complete clinical examination, biological tests (complete blood test) and a CT scan.

Follow-up period the completed treatment you will then be followed in consultation every 6 months for 2 years to evaluate the duration of the response to treatment and thus meet the objectives of the study.

ELIGIBILITY:
Inclusion Criteria:

* Immunophenotypically confirmed diagnosis of CLL (criteria iwCLL Hallek et al. 2018)
* Progressive CLL according to International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria
* Relapsed or refractory disease (≥ 1 previous line of treatment) with P53 genetic alteration (17p deletion and/or TP53 mutation).
* Age > 18 years
* Eastern Cooperative Oncology Group electrocorticogram (ECOG) status 0-2
* Negative serum pregnancy test one week prior to treatment for premenopausal women
* Cumulative Illness Rating Scale (CIRS) ≤ 6
* Life expectancy > 3 months.
* Possibility of follow-up
* Ability to understand the protocol
* Written informed consent of patient and treating physician

Exclusion Criteria:

* Previous treatment with ibrutinib.
* Patient refusal to perform bone marrow biopsy for evaluation point
* Prior other malignancy (except for adequately treated basal cell or squamous cell skin cancer, in situ cancer, or other cancer from which the subject has been disease free for ≥ 2 years).
* Known chronic obstructive pulmonary disease (COPD) with a Forced Expiratory Volume in 1 second (FEV1) < 50 % of predicted normal. FEV testing is required for patients suspected of having COPD.
* Moderate or severe persistent asthma within the two last years or currently uncontrolled asthma of any classification (American Lung Association criteria). Current controlled intermittent asthma or controlled mild persistent asthma is not an exclusion criterion.
* Patients with active bacterial, viral, or fungal infection requiring systemic treatment.
* Patients with known infection with human immunodeficiency virus (HIV) or human T-lymphotropic virus type 1 (HTLV-1)
* Active B or C hepatitis (positive Hepatitis B Virus surface antigen (HBsAg) or Hepatitis B Virus (HBV) DNA for HBV; Positive Hepatitis C virus (HCV) RNA for HCV)
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies.
* Any other uncontrolled medical condition or comorbidity that might interfere with subject's participation.
* Concomitant dual antiplatelet therapy
* Concomitant treatment with both antiplatelet and anticoagulation therapy
* Treatment with other investigational agent or participating to another trial within 30 days prior to entering the study
* Hemoglobin < 8 g/dL
* Absolute neutrophil count (ANC) < 1000/mm3
* Platelets < 30000/mm3
* Inadequate renal function: creatinine clearance < 50 ml/min (Cockcroft and Gault)
* Inadequate liver function: Aspartate Transaminase (ASAT), Alanine aminotransferase (ALT) > 2.5 x Upper Limit of Normal (ULN)
* Total bilirubin > 1.5 x ULN unless rise is due to Gilbert's syndrome or of non-hepatic origin.
* Active auto-immune haemolytic anemia
* Richter's transformation
* Evidence of central nervous system (CNS) involvement
* Pregnant or breastfeeding women.
* Adult under law-control
* Fertile male and female patients who cannot or do not wish to use an effective method of contraception, during and for 12 months after the final treatment used for the purposes of the study
* No affiliate to social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2023-06-17 (Actual); Study Completion 2025-12-19 (Estimated)

PRIMARY OUTCOMES:
Complete response rate (CR) at 12 months. | at 12 months
  Treatment response (ratio between the number of patients achieving complete response and the total number of patients included

SECONDARY OUTCOMES:
Occurrence of Tumor lysis syndrome | At the first infusion of daratumumab (day 1 and day 2) and at the second infusion of daratumumab (day 8)
  Frequency and severity of tumor lysis syndrome
Study treatment Emergent Adverse Events | From the first treatment administration and during treatment period (ibrutinib and daratumumab)
  Incidence and severity of study treatment-Emergent Adverse Events utilizing National Cancer Institute - Common Terminology Criteria (NCI-CTC) criteria v4.03.
Response rate | 12 months after beginning study treatment
  Overall response (OR) rate, partial response (PR) rate, PR with lymphocytosis rate
Minimal residual disease (MRD) assessement | During treatment :every 6 months after beginning study treatment until month 36 and 30 days after the last daratumumab infusion
  Presence of MRD measured by either quantitative PCR or flow cytometry
Progression Free Survival (PFS) | from date of inclusion to the date of first-documented progression, assessed up to 2 years
  time interval between the date of inclusion in the trial the date of progression of the illness or death
Overall Survival | from date of inclusion until the date of death, assessed up to 5 years
  time interval between the date of inclusion in the trial and the date of death
Duration of response | from the end of treatment to the date of progression, relapse or death, assessed up to 5 years
  time elapsed between the date of obtaining a maximal objective response (CR, PR or PR with persistent lymphocytosis) and the date of progression of the disease or death
CD38 expression in CLL cells | At baseline (day 0) and and before the first daratumumab perfusion (day 27)
  CD38 expression rate by immunophenotyping
Cumulative rate of Richter's syndrome | up to 5 years
  Number of patients who develop a Richter's syndrome

OTHER OUTCOMES:
Research of predictive biomarker and immune signatures in peripheral blood cells | At baseline and up to 3 years
  Deep phenotyping by high dimensional single cell mass cytometry (CyTOF) of peripheral blood cells

CONTACTS AND LOCATIONS:
Overall Officials: Alain DELMER, MD PD, Study Chair — French Innovative Leukemia Organisation; Thérèse AURRAN-SCHEINLITZ, MD, Principal Investigator — French Innovative Leukemia Organisation
Locations (24):
- France (24):
  - Chu Amiens Sud, Amiens
  - CH Annecy Genevois - Hématologie A3, Annecy
  - CHU Jean Minjoz - Hématologie, Besançon
  - Hôpital Avicenne - Centre de Recherche Clinique, Bobigny
  - CHU Caen - IHBN - Hématologie Clinique, Caen
  - CHU Estaing - Hématologie Clinique Adulte, Clermont-Ferrand
  - CHU Grenoble - Hématologie, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - Centre Hospitalier du Mans, Le Mans
  - Centre Léon Bérard - Hématologie, Lyon
  - CHLS - Lyon Pierre Bénite - Service Hématologie, Lyon
  - Institut Paoli-Calmettes - Hématologie Clinique, Marseille
  - Hôpital Saint-Eloi - Hématologie Clinique, Montpellier
  - CHU Hôtel Dieu - Hématologie Clinique, Nantes
  - Hôpital Pitié Salpétrière - Hématologie, Paris
  - CHU Bordeaux - Hôpital Haut-Lévèque - CFM Maladies du sang, Pessac
  - Hôpital de la Milétrie - Hématologie et Thérapie Cellulaire, Poitiers
  - Hôpital Robert Debré - Hématologie Clinique, Reims
  - CHU Pontchaillou - Hématologie Clinique BMT-HC, Rennes
  - Centre Henri Becquerel - Service Hématologie Clinique, Rouen
  - ICANS, Strasbourg
  - IUCT ONCOPOLE - Hématologie, Toulouse
  - Hôpital Bretonneau - Hématologie et Thérapie Cellulaire, Tours
  - Hôpitaux de Brabois - Hématologie Adulte, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: French Innovative Leukemia Organization (FILO) internet site — https://www.filo-leucemie.org/